CLINICAL TRIAL: NCT00577421
Title: An Extension Study to Assess BMD and Bone Turnover Response to 5 mg Daily Risedronate Treatment in Women With PMO
Brief Title: Study to Assess BMD and Bone Turnover Response to 5 mg Daily Risedronate Treatment in Women With PMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2002157
Record Dates: First submitted 2007-12-19; First posted 2007-12-20 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): 5 mg/day risedronate
  Interventions: Drug: risedronate

INTERVENTIONS:
Drug: risedronate — 5 mg tablet of risedronate once a day for 2 years

SUMMARY:
A 2-year, Multicenter, Open-label, Phase IIIb Extension Study to Assess Bone Mineral Density and Bone Turnover Response to 5 mg Daily Risedronate Treatment in Women with Postmenopausal Osteoporosis Who Sequentially Completed Clinical Studies RVE009093, RVE1996077, RVE1998080, and RVE2001079 (NCT01249261)

DETAILED DESCRIPTION:
A 2-year, Multicenter, Open-label, Phase IIIb Extension Study to Assess Bone Mineral Density and Bone Turnover Response to 5 mg Daily Risedronate Treatment in Women with Postmenopausal Osteoporosis Who Sequentially Completed Clinical Studies RVE009093, RVE1996077, RVE1998080, and RVE2001079 (NCT01249261)

ELIGIBILITY:
Inclusion Criteria:

* have satisfactorily completed Clinical Study RVE2001079 (Year 8 extension study)

Exclusion Criteria:

* Can not use any bone modifying substances except risedronate

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-06; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
To assess the safety and tolerability profile of 5 mg daily oral risedronate therapy administered for 2 years in patients with post-menopausal osteoporosis, who had received risedronate for 2 or 7 years and then had a risedronate-free year. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich H Wenderoth, MD, Study Director — Procter and Gamble
Locations (5):
- Research Site, Concord, Australia
- Research Facility, Siena, Italy
- Research Facility, Warsaw, Poland
- Research Facility, Barcelona, Spain
- Research Facility, Gothenburg, Sweden